CLINICAL TRIAL: NCT04466787
Title: Comparison of Spectral Photon Counting CT (SPCCT) With Dual Energy CT (DECT) and Magnetic Resonance Imaging (MRI) for Plaque and Lumen Carotid Arteries Evaluation.
Acronym: CAPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 69HCL18_0412; 2018-A02696-49 (Other: IDRCB)
Record Dates: First submitted 2020-03-19; First posted 2020-07-10 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Supra-Aortic Stenosis
Keywords: diagnostic; carotid plaque; SPCCT
MeSH Terms: conditions — Aortic Stenosis, Supravalvular; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The images will be read without knowing the CT scan used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spectral Photon Counting Computed Tomography (SPCCT) (Experimental): The randomized SPCCT patient will have this CT scan and an MRI before surgery. The plaque carotid will be collected for histological analysis
  Interventions: Diagnostic Test: Spectral Photon Counting Computed Tomography (SPCCT)
- Dual Energy CT (DECT) (Active Comparator): The randomized DECT patient will have this CT scan and an MRI before surgery. The plaque carotid will be collected for histological analysis
  Interventions: Diagnostic Test: Dual Energy CT (DECT)

INTERVENTIONS:
Diagnostic Test: Spectral Photon Counting Computed Tomography (SPCCT) — The acquisition for the assessment of the brain parenchyma and for the evaluation of the cervical and intracranial arteries will be performed without and with iodine based contrast media, respectively. The same parameters will be used for both conditions but for a large volume, from the aortic arch to the top of the head. The iodinate contrast agent's injection (Iomeron 400, Bracco Imaging France) will be performed at 5mL/s into an 18G catheter, followed by a 20 mL saline flush that will be injected at the same rate. The bolus volume will be determined according to the patient's body weight : 70 mL for patients < 80 kg and 1 mL/kg for patients > 80 kg, with a maximum of 90 mL.
  The SPCCT scanner is a prototype spectral photon-counting computed tomography system derived from a modified clinical CT system with a field of View (FOV) of 168 mm in-plane, and a z-coverage of 2 mm.
  Arms: Spectral Photon Counting Computed Tomography (SPCCT)
Diagnostic Test: Dual Energy CT (DECT) — The acquisition for the assessment of the brain parenchyma and for the evaluation of the cervical and intracranial arteries will be performed without and with iodine based contrast media, respectively. The same parameters will be used for both conditions but for a large volume, from the aortic arch to the top of the head. The iodinate contrast agent's injection (Iomeron 400, Bracco Imaging France) will be performed at 5mL/s into an 18G catheter, followed by a 20 mL saline flush that will be injected at the same rate. The bolus volume will be determined according to the patient's body weight : 70 mL for patients < 80 kg and 1 mL/kg for patients > 80 kg, with a maximum of 90 mL.
  DECT : IQon, Philips
  Arms: Dual Energy CT (DECT)

SUMMARY:
In this study, the investigator propose to determine the efficiency of a new and more sophisticated imaging prototype, the Spectral Photon Counting Computed Tomography (SPCCT), at characterizing vulnerable plaques and luminal stenosis in Carotid Atherosclerosis patients compared to DECT (Dual Energy CT) and MRI (Magnetic Resonance Imaging) which are used in current practice

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any ethnic background, aged > 18 years
* Any of the following known or suspected supra-aortic arterial disease based on : Prior stroke; Transient Ischemic Attack; Amaurosis Fugax; Referred for evaluation of any supra-aortic vessel; Follow-up for a stent in a supra-aortic vessel; Prior imaging ultrasounds study showing > ou = 50 % stenosis of a supra-aortic vessel segment (within 60 days before consent)
* Patient undergoing surgery within one month of carotid plaque evaluation
* Willingness and ability to follow directions and complete all study procedures specified in the protocol
* Pre-menopausal women only : Negative urinary pregnancy test on the day of imaging before the administration of study drug
* Patient has accepted to participate to the study and has signed the written consent
* Patient is affiliated to social security

Exclusion Criteria:

* Contraindication to MRI examinations (e.g. inability to hold breath, severe arrhythmias, very low cardiac output, severe claustrophobia, metallic devices not approved for MRI such as defibrillators, pacemaker, heart valve prostheses, cochlear implants, neuro-stimulators, implanted automated injection device, intraocular metallic foreign bodies, neurosurgical and vascular clips);
* Contraindication to the use of iodine and gadolinium containing contrast media (including subjects with suspicion for/or known to have NSF);- History of severe allergic or anaphylactic reaction to any allergen including drugs and contrast agents (as judged by the investigator, taking into account the intensity of the event);
* Estimated Glomerular Filtration Rate (eGFR) value < 30 mL/min/1.73 m2 derived from a serum creatinine result within 1 month before the imaging;
* Any subject on hemodialysis or peritoneal dialysis (Note: If there are multiple creatinine values, the values obtained prior to and closest to the time of the examination should be used);
* Acute renal insufficiency of any intensity, either due to hepato-renal syndrome or occurring in the per-operative liver transplantation period;
* Known subject history of severe cardiovascular disease (e.g. acute myocardial infarction [< 14 days], unstable angina, congestive heart failure New York Heart Association class IV) or known long QT syndrome;
* Suspected clinical instability or unpredictability of the clinical course during the study period (e.g. due to previous surgery);
* Scheduled or potentially expected for the period between the SPCCT or DECT and MRI: Any procedure that may alter the MRI or CT interpretation; Any interventional or surgical procedure involving the supra-aortic vessels.
* Pregnant or nursing (including pumping for storage and feeding); 11. Patient under guardianship, curators or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Lipid Necrotic Core (LNC) in mm² identified with SPCCT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Lipid Necrotic Core (LNC) in mm² identified with DECT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Lipid Necrotic Core (LNC) in mm² identified with histology | 1 month
  measurement of the height and thickness of surface of the plaque's components
Intra Plaque Hemorrhage (IPH) in mm² identified with SPCCT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Intra Plaque Hemorrhage (IPH) in mm² identified with DECT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Intra Plaque Hemorrhage (IPH) identified with histology | 1 month
  measurement of the height and thickness of surface of the plaque's components
Fibrous Cap Ulceration (FCU) in mm² identified with SPCCT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Fibrous Cap Ulceration (FCU) in mm² identified with DECT | 1 month
  measurement of the height and thickness of surface of the plaque's components
Fibrous Cap Ulceration (FCU) in mm² identified with histology | 1 month
  measurement of the height and thickness of surface of the plaque's components

SECONDARY OUTCOMES:
Number of irregularities identified with SPCCT | 1 month
  - Irregularities as defined by < 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Number of irregularities identified with DECT | 1 month
  - Irregularities as defined by < 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Number of irregularities identified with MRI | 1 month
  - Irregularities as defined by < 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Number of ulcerations identified with SPCCT | 1 month
  - Ulceration as defined by > 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Number of ulcerations identified with DECT | 1 month
  - Ulceration as defined by > 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Number of ulcerations identified with MRI | 1 month
  - Ulceration as defined by > 2 mm indentation, fissure, or erosion on the luminal surface of a plaque, exposing a portion of the inner plaque to direct contact with circulating blood.
Assessable vascular segments with lack of image artifacts | 1 month
  It will be assessed by estimating the image quality on scale from 1 to 4 (1 = poor, 2 = moderate, 3 = good, and 4 = excellent)
radiation dose received during SPCCT | 1 month
radiation dose received during DECT | 1 month
Tolerance to SPCCT assessed by a tolerance survey | 1 month
  1 to 10, 1= very bad, 10= very good. Survey adapted from Sparrow et al., Journal of magnetic resonance imaging 19:410-416, 2004
Tolerance to DECT assessed by a tolerance survey | 1 month
  1 to 10, 1= very bad, 10= very good. Survey adapted from Sparrow et al., Journal of magnetic resonance imaging 19:410-416, 2004
Tolerance to MRI assessed by a tolerance survey | 1 month
  1 to 10, 1= very bad, 10= very good. Survey adapted from Sparrow et al., Journal of magnetic resonance imaging 19:410-416, 2004

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DOUEK, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Louis Pradel cardiovascular Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided